CLINICAL TRIAL: NCT06998485
Title: Defining the Neurological Substrates of Proximal Upper Extremity Motor Control and Recovery After Stroke
Brief Title: Substrates for Post-Stroke Arm Rehabilitation
Acronym: SPARk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, David Lin, Neurologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025P000641; R01NS142153 (NIH)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Stroke Rehabilitation; Stroke; Neurorecovery
Keywords: stroke rehabilitation; motor control; neurorecovery; upper limb kinematics; corticospinal tract
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Mechanistic randomized controlled trial of arm basis training (a protocolized form of occupational therapy targeting proximal upper extremity motor control) versus usual care occupational therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Basis Training (Experimental): This program is a systematic training regimen specifically designed to improve proximal motor control for patients with severe upper extremity hemiparesis. The core principles of the Arm Basis Training Program focus on rebuilding the fundamental capacity for specific and selective motor control before progressing to more complex motor patterns.
  Interventions: Behavioral: Arm Basis Training
- Usual Care Occupational Therapy (No Intervention): Usual care occupational therapy. Participants will be asked to keep logs of the therapy they receive.

INTERVENTIONS:
Behavioral: Arm Basis Training — This program is a systematic training regimen specifically designed to improve proximal motor control for patients with severe upper extremity hemiparesis. The core principles of the Arm Basis Training Program focus on rebuilding the fundamental capacity for specific and selective motor control before progressing to more complex motor patterns.
  Arms: Arm Basis Training

SUMMARY:
Difficulty moving the arm is very common and a major cause of disability after stroke. Although rehabilitation therapies (i.e., occupational and physical therapy) are the most common treatments used to improve arm motor function, it remains unknown how therapy actually changes brain pathways after stroke. This project seeks to generate fundamental knowledge about brain pathways that allow people to move their arm after stroke and how these pathways change with rehabilitation; we expect this knowledge to translate to new therapies to reduce stroke-related disability.

We plan to enroll N = 50 patients with moderate to severe difficulty moving their arm after ischemic or hemorrhage stroke during the subacute period (3 to 6 months post stroke) into either 30 hours over 6 weeks of Arm Basis Training (a protocolized form of occupational therapy targeting motor control) or usual care. We will perform kinematic motor assessments, neuroimaging, and neurophysiology before and after therapy in order to test the hypothesis that intensive, target training improves arm motor control and induces corresponding anatomical and physiological changes of associated brain pathways.

DETAILED DESCRIPTION:
Strokes commonly damage motor pathways in the brain which leads to "hemiparesis", the collective term given to the syndrome of motor dysfunction after stroke. Upper extremity hemiparesis is comprised of both loss of abilities (negative signs- weakness and loss of dexterity or fractionated motor control) and intrusion of abnormal movements (positive signs- spasticity, abnormal resting postures, and synergies).

Recent work from our group and others shows that components of motor hemiparesis are dissociable: they can be separated and each map onto different and specific brain pathways. In this proposal, we focus on one specific component of post-stroke hemiparesis: proximal upper extremity motor control. Proximal upper extremity motor control can be measured as the ability to individuate and coordinate shoulder and elbow movements. We ask (i) where does proximal upper extremity motor control localize in the post-stroke brain? (ii) can we improve motor control with a specific form of targeted, high-dose, high-intensity therapy? And (iii) does therapy lead to corresponding changes in anatomy and physiology of brain pathways? Our central hypothesis is that intensive, targeted training improves proximal upper extremity motor control and induces corresponding anatomical and physiological changes of the corticospinal tract. To test this hypothesis, we will conduct three specific aims: (1) Determine baseline relationships between the corticospinal tract and proximal upper extremity motor control, (2) Define changes in proximal upper extremity motor control induced by targeted rehabilitation training, and (3) Define changes in corticospinal tract anatomy and physiology induced by targeted rehabilitation training. We leverage a clinical trial design of N = 50 patients with moderate-severe hemiparesis randomized to two groups: Arm Basis Training (a protocolized form of occupational therapy targeting motor control) versus usual care. Before and after six weeks of therapy, all patients will undergo kinematic assessment of motor control, diffusion magnetic resonance imaging to assess corticospinal tract axon density, and transcranial magnetic stimulation to assess corticospinal excitability. Dr. Lin, an acute care neurologist with neurorehabilitation and neuroscience training and the Director of the MGH Neurorecovery Clinic, will lead the project and bring together a world-class team of investigators and consultants, supported by the rich and multidisciplinary environment at Massachusetts General Hospital, Harvard Medical School, and collaborating institutions. This project is a mechanistic and hypothesis-driven investigation of the neuroanatomic and neurophysiologic signatures of a specific component of hemiparesis, proximal upper extremity motor control, and its response to targeted rehabilitation. The unique integration of kinematics, neuroanatomy, and neurophysiology in patients after stroke will transform stroke rehabilitation with a precision approach that targets brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

* first time unilateral ischemic or hemorrhagic stroke occurring within the 3-6 months
* upper extremity motor impairment as measured by the Upper Extremity Fugl-Meyer Assessment (UE-FMA) Score <= 44
* ability to participate in a 6-week intensive upper extremity intervention in English as determined by a licensed occupational therapist.

Exclusion Criteria:

* bilateral stroke
* unstable medical status affecting functional status
* pre-stroke upper extremity injury or conditions that limited use
* visual or auditory impairment limiting ability to participate in study procedures
* significant aphasia (NIHSS sub-item 9 > 1) or cognitive (NIHSS 1a or 1b or

  1c > 1) deficits
* known or expected inability to maintain follow-up through the study intervention and post- assessment
* contraindications to MRI
* contraindications to TMS
* known history of uncontrolled seizure disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Kinematic Measure of Upper Extremity Motor Control | Pre- and post- 6 weeks of therapy
  Kinematic measures of Upper Extremity Motor Control include joint individuation index (a measure of how well joints can move independently of other joints) and shoulder-elbow coordination (a measure of how normal a point-to-point planar reaching movement is)
Change in Corticospinal Tract Axon Density on MRI | Pre- and post- 6 weeks of therapy
  High-resolution diffusion MR neuroimaging will be performed, from which corticospinal tract axon density will be calculated
Change in Corticospinal Tract Neurophysiology | Pre- and post- six weeks of therapy
  The primary neurophysiologic measure of interest will be MEP presence or absence at proximal upper extremity muscles. If MEP positive, secondary measures of corticospinal excitability will be the MEP recruitment curve slope as well as MEP amplitude (at 100% MSO).

CONTACTS AND LOCATIONS:
Overall Officials: David J Lin, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
1. We will release raw behavior, imaging, and physiology data sets with relevant de-identified data to the database ~12 months after we have finished a portion of the project with enough sample size for publication. We will give database access to investigators who contact us about specific projects or analyses and/or are willing to enter into the same data sharing, authorship, and human subject data protection protocols that binds our multi-institutional collaboration, and agree to work closely with us to ensure that these complex data are analyzed with complete understanding of the experimental conditions under which they were collected.
  2. We will also release annotated, preprocessed datasets from this grant that form the basis for published manuscripts two years after their initial (online) publication date. We will make data available to individuals who agree to a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: May 2031 -
Access Criteria: We will give database access to investigators who contact us about specific projects or analyses and/or are willing to enter into the same data sharing, authorship, and human subject data protection protocols that binds our multi-institutional collaboration, and agree to work closely with us to ensure that these complex data are analyzed with complete understanding of the experimental conditions under which they were collected.